CLINICAL TRIAL: NCT00189007
Title: Does Antenatal Allopurinol Administration Reduce Post-hypoxic-ischemic Reperfusion Damage During Fetal Hypoxia in the Newborn?
Brief Title: Antenatal Allopurinol During Fetal Hypoxia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, dr. M.J.N.L. Benders, MD, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZonMw 170991001; ALLO-trial (Other: Dutch Consortium for Studies in Obstetrics and Gynaecology); 2006-005796-18 (EudraCT Number); 170991001 (Other Grant/Funding Number: ZonMw); NTR-1383 (Registry Identifier: Dutch Trial Register); NL26516.000.09 (Other: The Central Committee on Research Involving Human Subjects (CCMO))
Record Dates: First submitted 2005-09-11; First posted 2005-09-16 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Fetal Hypoxia; Reperfusion Injury
Keywords: allopurinol; neuroprotection; reperfusion injury; fetal hypoxia; post hypoxic-ischemic reperfusion damage
MeSH Terms: conditions — Fetal Hypoxia; Reperfusion Injury | interventions — Allopurinol; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Experimental): 500 mg allopurinol/ 50 mL water for injection intravenously
  Interventions: Drug: Allopurinol sodium
- Placebo (Placebo Comparator): 500 mg mannitol/50 mL water for injection intravenously
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Allopurinol sodium — Allopurinol sodium 500 mg / 50 mL, intravenously, single dose
  Other Names: Acepurin
  Arms: Allopurinol
Drug: Mannitol — Mannitol 500 mg/50 mL water for injection, intravenously, single dose
  Arms: Placebo

SUMMARY:
A former study (submitted) in 32 severely asphyxiated infants participating in a randomized double blind study, in which early postnatal allopurinol or a placebo (within 4 hours after birth) was administered to reduce free radical formation and consequently reperfusion/reoxygenation injury to the newborn brain, showed an unaltered high mortality and no clinically relevant improvement in morbidity in infants treated with allopurinol. It was hypothesized that postnatal allopurinol treatment started too late to reduce reperfusion-induced free radical surge and that initiating allopurinol treatment of the fetus with (imminent) hypoxia already via the mother during labor will be more effective to reduce free radical-induced post-asphyxial brain damage.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 36 weeks or more
* Non-reassuring CTG, significant events on the STAN-monitor AND/OR FBS < 7.20

Exclusion Criteria:

* Chromosomal abnormalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Free radical production and markers of neuronal damage | Up to 24 hours postpartum

SECONDARY OUTCOMES:
Developmental outcome | Up to 5 years of age
Mortality | Up to 28 days postpartum
Severe composite morbidity | Up to 28 days postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Frank van Bel, Prof MD PhD, Study Director — Wilhelmina Children's Hospital/UMC Utrecht; Manon JN Benders, MD, PhD, Principal Investigator — UMC Utrecht; Jan B Derks, MD, PhD, Principal Investigator — UMC Utrecht; Joepe J Kaandorp, MD, Principal Investigator — UMC Utrecht; Gerard H Visser, MD, PhD, Principal Investigator — UMC Utrecht; Ben WJ Mol, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Carin MA Rademaker, PhD, Principal Investigator — Clinical Pharmacy, UMCU
Locations (11):
- Netherlands (11):
  - Wilhelmina Children's Hospital/UMC Utrecht, Utrecht, Utrecht
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - AMC, Amsterdam
  - VUmc, Amsterdam
  - Gelre hospitals, Apeldoorn
  - Groene Hart Hospital, Gouda
  - UMCG, Groningen
  - LUMC, Leiden
  - Maastricht University Medical Center, Maastricht
  - Diakonessenhuis, Utrecht
  - Maxima Medical Center, Veldhoven

REFERENCES:
- [Background] Kaandorp JJ, Benders MJ, Rademaker CM, Torrance HL, Oudijk MA, de Haan TR, Bloemenkamp KW, Rijken M, van Pampus MG, Bos AF, Porath MM, Oetomo SB, Willekes C, Gavilanes AW, Wouters MG, van Elburg RM, Huisjes AJ, Bakker SC, van Meir CA, von Lindern J, Boon J, de Boer IP, Rijnders RJ, Jacobs CJ, Uiterwaal CS, Mol BW, Visser GH, van Bel F, Derks JB. Antenatal allopurinol for reduction of birth asphyxia induced brain damage (ALLO-Trial); a randomized double blind placebo controlled multicenter study. BMC Pregnancy Childbirth. 2010 Feb 18;10:8. doi: 10.1186/1471-2393-10-8. PMID 20167117
- [Derived] Klumper J, Kaandorp JJ, Schuit E, Groenendaal F, Koopman-Esseboom C, Mulder EJH, Van Bel F, Benders MJNL, Mol BWJ, van Elburg RM, Bos AF, Derks JB; ALLO-trial study group. Behavioral and neurodevelopmental outcome of children after maternal allopurinol administration during suspected fetal hypoxia: 5-year follow up of the ALLO-trial. PLoS One. 2018 Aug 23;13(8):e0201063. doi: 10.1371/journal.pone.0201063. eCollection 2018. PMID 30138355
- [Derived] Kaandorp JJ, Benders MJ, Schuit E, Rademaker CM, Oudijk MA, Porath MM, Oetomo SB, Wouters MG, van Elburg RM, Franssen MT, Bos AF, de Haan TR, Boon J, de Boer IP, Rijnders RJ, Jacobs CJ, Scheepers LH, Gavilanes DA, Bloemenkamp KW, Rijken M, van Meir CA, von Lindern JS, Huisjes AJ, Bakker SC, Mol BW, Visser GH, Van Bel F, Derks JB. Maternal allopurinol administration during suspected fetal hypoxia: a novel neuroprotective intervention? A multicentre randomised placebo controlled trial. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F216-23. doi: 10.1136/archdischild-2014-306769. Epub 2014 Dec 15. PMID 25512466
- [Derived] Kaandorp JJ, van den Broek MP, Benders MJ, Oudijk MA, Porath MM, Bambang Oetomo S, Wouters MG, van Elburg R, Franssen MT, Bos AF, Mol BW, Visser GH, van Bel F, Rademaker CM, Derks JB; ALLO-trial Study Group. Rapid target allopurinol concentrations in the hypoxic fetus after maternal administration during labour. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F144-8. doi: 10.1136/archdischild-2013-304876. Epub 2013 Dec 18. PMID 24352085
- [Derived] Torrance HL, Benders MJ, Derks JB, Rademaker CM, Bos AF, Van Den Berg P, Longini M, Buonocore G, Venegas M, Baquero H, Visser GH, Van Bel F. Maternal allopurinol during fetal hypoxia lowers cord blood levels of the brain injury marker S-100B. Pediatrics. 2009 Jul;124(1):350-7. doi: 10.1542/peds.2008-2228. PMID 19564319